CLINICAL TRIAL: NCT02738177
Title: Misoprostol Versus Effox (Individually or in Combination) as Cervical Ripening Agent Prior to 1st Trimesteric Surgical Evacuation
Brief Title: Misoprostol Versus Effox as Cervical Ripening Agent Prior Surgical Evacuation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moutaz Sherbini, lecturer of obs& gyn, Cairo University
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: 17480
Record Dates: First submitted 2016-04-09; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Ripening
Keywords: misopristol; effox; cervical ripening
MeSH Terms: interventions — Misoprostol; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- misoprostol group (Active Comparator): 30 candidates were receive 2 tablets of misoprostol (PGE1) 200ug (i.e. 400 ug) 4 hrs prior to surgical evacuation
  Interventions: Drug: Misoprostol
- Effox group (Active Comparator): 30 candidates were received 2 tablets of Effox (Isosorbide mononitrate) 20 mg (i.e 40 mg) 4 hrs prior to surgical evacuation
  Interventions: Drug: Isosorbide-5-mononitrate
- combination therapy group (Active Comparator): 30 candidates were received 1 tablets of misoprostol 200ug & 1 tablets of Effox 20 mg 4 hrs prior to surgical evacuation.
  Interventions: Drug: misoprostol and Isosorbide-5-mononitrate

INTERVENTIONS:
Drug: Misoprostol — 2 tablets of misoprostol (i.e. 400 ug) 4 hrs prior to surgical evacuation high up in the posterior fornix (misoprostol group)
  Other Names: mesotac; cytotec
  Arms: misoprostol group
Drug: Isosorbide-5-mononitrate — 2 tablets of Effox (i.e. 40 mg) 4 hrs prior to surgical evacuation high up in the posterior fornix (effox group)
  Other Names: Effox
  Arms: Effox group
Drug: misoprostol and Isosorbide-5-mononitrate — 1tablets of misoprostol (i.e.200 ug) & 1 tablets of Effox (i.e. 20 mg) 4 hrs prior to surgical evacuation high up in the posterior fornix (combination therapy group)
  Arms: combination therapy group

SUMMARY:
Ninety healthy pregnant women candidate for surgical evacuation after confirming 1st trimester pregnancy loss were enrolled in the study. They were randomized in three groups; misoprostol group in which 30 candidates were receive 2 tablets of misoprostol (i.e. 400 ug) 4 hrs prior to surgical evacuation, Effox group in which 30 candidates were received 2 tablets of Effox (i.e 40 mg) 4 hrs prior to surgical evacuation & combination therapy group in which 30 candidates were received 1 tablets of misoprostol 200ug & 1 tablets of Effox 20 mg 4 hrs prior to surgical evacuation. For all participants, the route of administration was the intravaginal route 1ry outcomes included cervical consistency & dilatation immediately before the procedure. 2ry outcomes included total duration of the operation and the occurrence of drug-related side effects

DETAILED DESCRIPTION:
Objective: To compare the efficacy of the individual use of Misoprostol or Effox or their combination as cervical ripening agents in cases with 1st trimesteric pregnancy loss candidate for surgical evacuation.

Study Design: A randomized Single-blind comparative study. Setting: The Obstetrics and Gynecology casuality department of Kasr El Aini hospital (Cairo University - Egypt) in the period from November 2015 to June 2016.

Methodology: ninety healthy pregnant women candidate for surgical evacuation after confirming 1st trimester pregnancy loss were enrolled in the study. They were randomized in three groups; misoprostol group in which 30 candidates were receive 2 tablets of misoprostol (PGE1) 200ug (i.e. 400 ug) 4 hrs prior to surgical evacuation, Effox group in which 30 candidates were received 2 tablets of Effox (Isosorbide mononitrate) 20 mg (i.e 40 mg) 4 hrs prior to surgical evacuation & combination therapy group in which 30 candidates were received 1 tablets of misoprostol 200ug & 1 tablets of Effox 20 mg 4 hrs prior to surgical evacuation. The study was approved by the Hospital Ethical Committee. Informed consents were obtained from all participants after explanation of the aim of the study & the potential adverse effects. The study was not supported by any pharmacological company.

Inclusion criteria included maternal age 18-40 years, 1st trimesteric pregnancy loss with gestational age 12 weeks or less (diagnosis was confirmed using transvaginal ultrasound according to the following criteria: Crown-rump length {CRL} of 7 mm or more and no heartbeat, Mean sac diameter {MSD} of 25 mm or more and no embryo, absence of embryo with heartbeat 2 wk or more after a scan that showed a gestational sac without a yolk sac and absence of embryo with heartbeat 11 days or more after a scan that showed a gestational sac with a yolk sac)* & closed firm cervix. Exclusion criteria included evidence suggesting spontaneous onset of abortion (vaginal bleeding or and uterine cramps), previous trial to induce abortion or the use of any cervical ripening agent during the current pregnancy, presence or suspicion of septic abortion (fever > 38 C, offensive vaginal discharge & leukocytosis), Uterine anomalies or history of any cervical surgery or manipulation. For all patients, full history was taken followed by complete physical examination (including cervical assessment), transvaginal ultrasound (to confirm early pregnancy loss) & routine preoperative investigation. Patient is then randomized to one of the three groups (using computer generated random numbers) and accordingly the investigator gave her either 2 tablets of misoprostol 200ug (misoprostol group) or 2 tablets of Effox 20 mg (Effox group) or 1 tablets of misoprostol 200ug & 1 tablets of Effox 20 mg (Combination therapy group). For all participants, the route of administration was the intravaginal route (tablets were places high up in the posterior fornix of the vagina. Only patients were blinded to the nature of the tablets. 4 hrs later, the patient was admitted to the operating room for surgical evacuation with the following technique: under general anesthesia & after assessment of cervical consistency (soft or firm) & dilatation (tested by the number of the largest Hegar's dilator passed without resistance), ultrasound-guided suction evacuation was done followed by fine curettage using the appropriate size curette. All participants were monitored for any changes in vital signs (every hour), occurrence of headache & severe abdominal cramps since the onset of drug administration till 6 hours postoperative. 1ry outcomes included cervical consistency & dilatation immediately before the procedure. 2ry outcomes included total duration of the operation and the occurrence of drug-related side effects namely high temperature (38 or more) and severe abdominal pain for the misoprostol or headache and low blood pressure for the Effox.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women candidate for surgical evacuation
* 1st trimesteric pregnancy loss with gestational age 12 weeks or less (diagnosis was confirmed using transvaginal ultrasound according to the following criteria: Crown-rump length {CRL} of 7 mm or more and no heartbeat, Mean sac diameter {MSD} of 25 mm or more and no embryo, absence of embryo with heartbeat 2 wk or more after a scan that showed a gestational sac without a yolk sac and absence of embryo with heartbeat 11 days or more after a scan that showed a gestational sac with a yolk sac)
* closed and firm cervix

Exclusion Criteria:

* evidence suggesting spontaneous onset of abortion (vaginal bleeding or and uterine cramps), previous trial to induce abortion or the use of any cervical ripening agent during the current pregnancy, presence or suspicion of septic abortion (fever > 38 degree Centigrade, offensive vaginal discharge & leukocytosis), Uterine anomalies or history of any cervical surgery or manipulation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
cervical dilatation | 4 hours after receiving the drug
  tested by the number of the largest Hegar's dilator passed without resistance

SECONDARY OUTCOMES:
misoprostol side effects | since receiving the drug till 6 hours postoperative
  high temperature (38 degree centigrade or more) and severe abdominal pain.
effox side effects | since receiving the drug till 6 hours postoperative
  headache and low blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Moutaz Elsherbini, MD, Principal Investigator — Lecturer of obs & gyn
Locations (1):
- Kasr Elainy Hospital (Cairo University), Cairo, Cairo Governorate, Egypt